CLINICAL TRIAL: NCT00000705
Title: A Phase I Trial to Evaluate Azidothymidine (AZT) in the Treatment of HIV Infections in Patients With Hemophilia
Brief Title: Safety and Effectiveness of Azidothymidine (AZT) in HIV-Positive Patients With Hemophilia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 017; 10993 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hemophilia A
Keywords: Drug Evaluation; Zidovudine; Hemophilia A
MeSH Terms: conditions — HIV Infections; Hemophilia A | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see if giving azidothymidine (AZT) to HIV-positive patients with hemophilia is safe and if it is effective in lowering HIV levels and boosting the immune system.

HIV infects and inactivates certain blood cells that are part of the body's immune system. The damage to the body's immune system can result in unusual infections and/or unusual forms of cancer. A large percentage of hemophiliacs are HIV-positive and there is a clear risk for the development of AIDS in these patients. AZT may be effective in lowering HIV levels and boosting the immune system but its side effects are not understood in these patients.

DETAILED DESCRIPTION:
There is a clear risk for development of AIDS in hemophilic patients. AZT administration has been shown to inhibit HIV replication in vitro. Patients taking AZT have experienced fewer opportunistic infections and improvements in measures of immunity. The most common laboratory abnormalities observed with AZT are hematologic. However, the clinical and laboratory toxicity of AZT remains poorly understood in hemophiliacs. Hepatitis and liver dysfunction are more common in this population compared to other groups at risk for HIV infection. Because AZT is largely metabolized in the liver, drug pharmacokinetics needs to be evaluated in this patient population.

Both hemophiliacs and non-hemophiliacs take AZT for a period of 12 weeks. The first dose is administered intravenously. AZT is then given orally every 4 hours while awake (5 doses per day). Patients are evaluated by physical examinations and laboratory assessments. These include HIV culture of blood and leukocyte counts, lymphocyte counts, and lymphocyte subsets measured at study entry and every 4 weeks thereafter. Patients are hospitalized for pharmacokinetic studies at study entry and at Weeks 6 and 12. Each of these studies involves both intravenous and oral administration within 48 hours of one another. Blood is sampled at 0, 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours after each administration and urine is collected every 2 hours for 12 hours.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a bleeding disorder such as hemophilia A or B, a lack of factor VIII (a blood clotting factor), or severe von Willebrand's disease.
* Will be available for follow-up for at least a year.
* Are at least 12 years old (consent of parent or guardian required if under 18).
* Are willing to use an effective method of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a life-threatening opportunistic (AIDS-related) infection or AIDS-related symptoms.
* Have taken certain drugs within 30 days prior to study entry including chemotherapy and interferon.
* Are taking acetaminophen or drugs containing acetaminophen.
* Are pregnant or breast-feeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Study Completion 1989-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Reichman, Study Chair
Locations (2):
- United States (2):
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Univ of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Background] Portmore A, Morse G, Hewitt R, Reichman R. Comparative oral disposition of zidovudine in neutropenic AIDS patients and asymptomatic hemophiliacs. Int Conf AIDS. 1990 Jun 20-23;6(3):196 (abstract no SB442)
- [Background] Morse GD, Portmore A, Olson J, Taylor C, Plank C, Reichman RC. Multiple-dose pharmacokinetics of oral zidovudine in hemophilia patients with human immunodeficiency virus infection. Antimicrob Agents Chemother. 1990 Mar;34(3):394-7. doi: 10.1128/AAC.34.3.394. PMID 2334151
- [Background] Morse GD, Olson J, Portmore A, Taylor C, Plank C, Reichman RC. Pharmacokinetics of orally administered zidovudine among patients with hemophilia and asymptomatic human immunodeficiency virus (HIV) infection. Antiviral Res. 1989 Mar;11(2):57-65. doi: 10.1016/0166-3542(89)90008-9. PMID 2729955
- [Background] Morse G, Olson J, Portmore A, Taylor C, Plank C, Reichman R. Intravenous and oral pharmacokinetics of zidovudine in hemophilia patients with human immunodeficiency virus infection. Int Conf AIDS. 1989 Jun 4-9;5:278 (abstract no MBP342)